CLINICAL TRIAL: NCT00558753
Title: A Prospective, Randomized Controlled Trial on Perioperative Pregabalin to Reduce Late-onset Complex Regional Pain Syndrome After Total Knee Arthroplasty
Brief Title: Prospective, Randomized Controlled Trial on Perioperative Pregabalin to Reduce Late-onset CRPS After TKA
Acronym: PregTKA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Asokumar Buvanendran, Attending Physician, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABuv102007
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: CRPS
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Placebo (Placebo Comparator): Half of the patients will receive PO placebo for 14 days
  Interventions: Drug: Placebo
- 2 Pregabalin (Experimental): PO pregabalin 300 mg 2 hours prior to surgery, and 150 mg twice a day for 10 postoperative days. Pregabalin will be tapered to 75 mg twice daily between days 11 to 12 and then to 50 mg twice daily between days 13 to 14 post operatively and then stopped.
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — PO pregabalin 300 mg 2 hours prior to surgery, and 150 mg twice a day for 10 postoperative days. Pregabalin will be tapered to 75 mg twice daily between days 11 to 12 and then to 50 mg twice daily between days 13 to 14 post operatively and then stopped.
  Other Names: Lyrica
  Arms: 2 Pregabalin
Drug: Placebo — Placebo for Given 2 hours prior to surgery, and twice a day for 14 postoperative days.
  Arms: 1 Placebo

SUMMARY:
The Department of Anesthesiology is conducting a clinical trial to evaluate if pregabalin given prior to and for several days after Total Knee Arthroplasty (TKA) will reduce the prevalence of Complex Regional Pain Syndrome (CRPS) at late postoperative times. The prevalence of complex regional pain syndrome (CRPS) following total knee arthroplasty (TKA) is 13% at 6 months post-surgery. CRPS is a painful debilitating condition, with 4 main classes of symptoms : sensory, including burning, allodynia, and hyperalgesia in the affected limb; vasomotor, including temperature asymmetry and skin color changes; edema and sudomotor, including sweating; and movement disorders and dystrophy, including decreased range of motion, motor dysfunction (weakness, tremor, dystonia) and changes in hair, nails or skin.

DETAILED DESCRIPTION:
The Department of Anesthesiology is conducting a clinical trial to evaluate if pregabalin given prior to and for several days after Total Knee Arthroplasty (TKA) will reduce the prevalence of Complex Regional Pain Syndrome (CRPS) at late postoperative times. The prevalence of complex regional pain syndrome (CRPS) following total knee arthroplasty (TKA) is 13% at 6 months post-surgery. CRPS is a painful debilitating condition, with 4 main classes of symptoms : sensory, including burning, allodynia, and hyperalgesia in the affected limb; vasomotor, including temperature asymmetry and skin color changes; edema and sudomotor, including sweating; and movement disorders and dystrophy, including decreased range of motion, motor dysfunction (weakness, tremor, dystonia) and changes in hair, nails or skin.

Gabapentin and the related more potent compound pregabalin have been shown to reduce postoperative pain in animal models. Pregabalin also reduces neuropathic pain in rats. In patients, gabapentin has been administered before surgery to treat postoperative pain. In addition, pregabalin has been given postoperatively to reduce dental pain after molar extraction. Gabapentin has been used for many years in patients with neuropathic pain, including reflex sympathetic dystrophy. More recently, pregabalin has also been shown to be efficacious in the treatment of neuropathic pain. However, no clinical study has investigated whether perioperative administration of gabapentin or pregabalin can reduce persistent long-term pain syndromes e.g. CRPS.Subjects between the ages of 21 and 80 will be recruited after obtaining an Informed Consent.

ELIGIBILITY:
Inclusion Criteria:

1. History of osteoarthritis
2. Subjects who can understand and communicate in English.

Exclusion Criteria:

1. Younger than 21 years or older than 80 years.
2. American Society of Anesthesiologists physical status IV.
3. Prior usage of gabapentin (or pregabalin) will not be an exclusionary criterion; however, patients will have been withdrawn from these medications for at least 7 days before surgery.
4. Patients with a history of neuropathic pain conditions.
5. Patients who are currently enrolled in another investigational study.
6. Pre-existing heart conditions
7. Patients on thiazolidinedione class of anti-diabetic medications (eg. rosiglitazone, pioglitazone).

   -

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, M.D., Principal Investigator — Rush University Medical Center

REFERENCES:
- [Result] Buvanendran A, Kroin JS, Della Valle CJ, Kari M, Moric M, Tuman KJ. Perioperative oral pregabalin reduces chronic pain after total knee arthroplasty: a prospective, randomized, controlled trial. Anesth Analg. 2010 Jan 1;110(1):199-207. doi: 10.1213/ANE.0b013e3181c4273a. Epub 2009 Nov 12. PMID 19910619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 2006 to August 2007, 350 consecutive patients scheduled to undergo elective primary Total knee arthroplasty (TKA) were contacted and assessed for study eligibility. There were 110 Screen Failures (31 Not meeting inclusion criteria, 79 eligible but did not give consent), resulting in 240 enrolled subjects.
Pre-assignment Details: There were 110 Screen Failures (31 Not meeting inclusion criteria, 79 eligible but did not give consent), resulting in 240 enrolled subjects.
Groups:
- 1 Placebo: Half of the patients will receive oral (PO) placebo for 14 days
Period: Overall Study
Arm/Group | 1 Placebo | 2 Pregabalin
Started | 120 | 120
Completed | 115 | 113
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Placebo | 2 Pregabalin | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.9) | 64.0 (8.3) | 63.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 91 | 175
  Male | 36 | 29 | 65
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index...........................................
  kg/m^2 | 34.6 (7.7) | 34.2 (8.4) | 34.4 (8)

OUTCOME MEASURES:

1. Primary Outcome: Epidural Medication Consumption Rate
Description: Epidural medication consumption was recorded for each 4-h interval from the completion of surgery to the time that the epidural was discontinued (same as the time to achieve hospital discharge criteria). Because the discontinuation time varied from patient to patient (as they achieved physical therapy criteria), the average hourly consumption (total analgesic used divided by the total infusion time) was used as the measure of epidural drug use.
Time Frame: 36 h
Population: Because of structural missing data, sample sizes are smaller than the samples size for the secondary measure.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | 1 Placebo | 2 Pregabalin
Number analyzed (Participants) | 76 | 70
mL/h | 6.40 (1.26) | 5.77 (1.31)
Statistical Analysis 1: Comparison: 1 Placebo vs 2 Pregabalin; Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = 0.63

2. Secondary Outcome: Neuropathic Pain (S-LANSS > 12)
Description: Patients will be evaluated in blinded fashion for lower extremity Complex Regional Pain Syndrome(CRPS) at pre-op, 1, 3, and 6 months postsurgery based initially on telephone interviews. An S-LANSS score of 12 or more was an indication of chronic neuropathic pain. Patients with an Self-report version of the Leeds Assessment of Neuropathic Symptoms and Signs(S-LANSS) score of 12 or more at 6 mo came to the physician's office for a standardized physical examination, which included the S-LANSS examination items (allodynia and hyperalgesia) directly assessed by the physician, plus a pinprick evaluation.
Time Frame: 3 and 6 months post-surgery
Measure: Number; unit: participants
Arm/Group | 1 Placebo | 2 Pregabalin
Number analyzed (Participants) | 115 | 113
participants
  Neuropathic pain at 3 Month Follow up | 10 | 0
  Neuropathic pain at 6 Month Follow up | 6 | 0
Statistical Analysis 1: Comparison: 1 Placebo vs 2 Pregabalin; For 3 month followup on incidence of neuropathic pain; Test type: Superiority or Other; p = 0.0013, Chi-squared; Independence: Chi-squared = 10.3
Statistical Analysis 2: Comparison: 1 Placebo vs 2 Pregabalin; For 6 month followup on incidence of neuropathic pain; Test type: Superiority or Other; p = 0.0139, Chi-squared; Independence: Chi-squared = 6.05

3. Secondary Outcome: Knee Range of Motion (Active Flexion)
Time Frame: 1-30 days
Measure: Least Squares Mean (Standard Error); unit: Degrees
Arm/Group | 1 Placebo | 2 Pregabalin
Number analyzed (Participants) | 89 | 73
Degrees
  Day 1 | 75.6 (1.5) | 77.8 (1.6)
  Day 2 | 76.7 (1.3) | 81.0 (1.4)
  Day 3 | 80.4 (1.5) | 84.2 (1.6)
  Day 30 | 103.0 (1.3) | 107.2 (1.4)
Statistical Analysis 1: Comparison: 1 Placebo vs 2 Pregabalin; Mixed model test of condition (Placebo v Pregabalin) main effect; Test type: Superiority or Other; p = 0.0133, Mixed Models Analysis — Test of condition(Placebo v Pregabalin) main effect; Mixed model with main effects and time by condition interaction; Slope = -4.2
Statistical Analysis 2: Comparison: 1 Placebo vs 2 Pregabalin; Test of Condition Effect (Placebo v Pregabalin) at the 1-day post surgery time point (Slice); Test type: Superiority or Other; p = 0.3097, Mixed Models Analysis; Mixed model test of Condition Effect (Placebo v Pregabalin) at the 1-day post surgery time point (Slice); Interaction Slice F-value = 1.04
Statistical Analysis 3: Comparison: 1 Placebo vs 2 Pregabalin; Test of Condition Effect (Placebo v Pregabalin) at the 2-day post surgery time point (Slice); Test type: Superiority or Other; p = 0.0247, Mixed Models Analysis; Interaction Slice F-value = 5.10
Statistical Analysis 4: Comparison: 1 Placebo vs 2 Pregabalin; Test of Condition Effect (Placebo v Pregabalin) at the 3-day post surgery time point (Slice); Test type: Superiority or Other; p = 0.0786, Mixed Models Analysis; Interaction Slice F-value = 3.11
Statistical Analysis 5: Comparison: 1 Placebo vs 2 Pregabalin; Test of Condition Effect (Placebo v Pregabalin) at the 30-day post surgery time point (Slice); Test type: Superiority or Other; p = 0.0254, Mixed Models Analysis; Interaction Slice F-value = 5.04

ADVERSE EVENTS:
Arm/Group | 1 Placebo | 2 Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 65/120 | 69/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Placebo (N=120) | 2 Pregabalin (N=120)
Sedation (General disorders) | 28 | 35
Confusion (Gastrointestinal disorders) | 9 | 15
Dizziness (General disorders) | 16 | 25
Headache (Gastrointestinal disorders) | 0 | 3
Dry Mouth (General disorders) | 3 | 9
Nausea (General disorders) | 27 | 17
Vomiting (General disorders) | 10 | 9
Itching (General disorders) | 13 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes